CLINICAL TRIAL: NCT06080945
Title: Tailored Pharmacist-led Intervention to Improve Adherence to Budesonide in Asthmatic Children
Brief Title: Tailored Pharmacist-led Intervention to Improve Adherence to Budesonide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaoxing Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Xu Renjie, Principal Investigator, Shaoxing Maternity and Child Health Care Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ShaoxingMaternityChild
Record Dates: First submitted 2023-09-20; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-led care group (Experimental): In addition to usual care, the patient in the intervention group received pharmacist-led multidisciplinary care. The multidisciplinary team consists of a physician, a pharmacist and a nurse. To ensure the uniformity of the material provided during counseling sessions, all professionals attended training before beginning to work with patients. Patients in the control group were given the hospital's standard of care discharge counseling on budesonide, whereas patients in the intervention group were given both the standard of care counseling and a pharmacist-driven discharge counseling on budesonide. A pharmacist first spoke with the parents to obtain comprehensive medical, familial, and social histories. After personalized pharmacogenetic testing, a pamphlet with instructions on how to take their medications was given to each parent.
  Interventions: Other: pharmacist-led patient-centered medication therapy management
- Usual care group (No Intervention): The control group will receive care as usual

INTERVENTIONS:
Other: pharmacist-led patient-centered medication therapy management — The intervention group will receive a pharmacist-driven discharge counseling on budesonide, an inhaled glucocorticoid, from recruitment, until 12 months.
  Arms: Pharmacist-led care group

SUMMARY:
Gaining control of asthma can be especially difficult during childhood as children undergo a variety of biological, developmental, and psychosocial changes. This study was designed to evaluate the impact of a pharmacist-led patient-centered medication therapy management trial on asthma and medication adherence among children receiving budesonide at a tertiary hospital in Shaoxing, China. In this randomised controlled trial, one hundred and two children, with asthma, from 6 to 14 age, will be recruited and randomised to an intervention group or a control group. The intervention group will receive a pharmacist-driven discharge counseling on budesonide, an inhaled glucocorticoid, from recruitment, until 12 months. The control group will receive care as usual. The main outcomes were spirometry measurements and medication adherence estimation.

DETAILED DESCRIPTION:
The patient in the intervention group received pharmacist-led multidisciplinary care. The multidisciplinary team consists of a physician, a pharmacist and a nurse. To ensure the uniformity of the material provided during counseling sessions, all professionals attended training before beginning to work with patients. Patients in the control group were given the hospital's standard of care discharge counseling on budesonide, whereas patients in the intervention group were given both the standard of care counseling and a pharmacist-driven discharge counseling on budesonide. A pharmacist first spoke with the parents to obtain comprehensive medical, familial, and social histories. After personalized pharmacogenetic testing, a pamphlet with instructions on how to take their medications was given to each parent . Then, they were provided with an educational pamphlet during discharge, Parents signed in the educational pamphlet to confirm that they had received the medication information . The pamphlet contained general advice on lifestyle changes while taking budesonide, how to handle gastrointestinal reactions if it occurs, general safety measures, and details on over-the-counter medications that might interact with inhaled corticosteroid (ICS). The pamphlet included details on how often to take the medication, management about missing doses, how to store it, how food and medications interact with it, and any other information relevant to budesonide. Pharmacists explained the content of the pamphlet to the parents, and answered any question related to the drug. All parents in the pharmacist-led group got phone calls from pharmacists as part of the routine clinical follow-up to evaluate their use of ICS, to clarify any uncertainties, and to contact their doctors as necessary to address any problems that were discovered. At intervals of one to three months, in conjunction with the dates for clinical follow-up appointments or medication refills, the parents were informed of planned follow-up conversations over the phone or in person. Each visit included a planned, one-on-one education session on medications.

ELIGIBILITY:
Inclusion Criteria:

* 6-14 years-of-age
* Met the diagnostic criteria described by the "Recommendations for Standardized Diagnosis and Treatment of Bronchial Asthma in Children (2020 Edition)"
* Dysfunctional lung function with a positive provocation test
* No previous respiratory rehabilitation treatment
* The parents' written informed consent.

Exclusion Criteria:

* Acute exacerbation of asthma
* The co-existence of other respiratory system diseases (such as bronchopneumonia and bronchopulmonary dysplasia), cardiovascular system diseases (myocarditis and congenital heart disease), motor nervous system diseases
* The presence of mental disorders or the patient had psychological abnormalities and could not cooperate.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-11-08 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Spirometry Measurements | during the intervention (up to 1 year)
  Spirometry measurements was measured using a lung function tester (JAEGER, Germany). Measurement indicators were shown as forced expiratory volume in one second (FEV1). The percentage (%) of the actual value to the expected value was used for data analysis.
Medication adherence assessment | during the intervention (up to 1 year)
  Previous studies show medication adherence estimation and differentiation scale (MEDS) has proven good reliability and validity . The MEDS version had 16 items, and each "Never" response received a score of "1," "Rarely" received a score of "2," "Sometimes" received a score of "3," "Often" received a score of "4", and "Always" received a score of "5". Consequently, a patient could receive an overall number between 16 (perfectly adherent) and 80 (completely non-adherent).

CONTACTS AND LOCATIONS:
Overall Officials: Renjie Xu, Principal Investigator — Shaoxing Maternity and Child Health Care Hospital
Locations (1):
- Shaoxing Maternity and Child Care hospital, Shaoxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No